CLINICAL TRIAL: NCT07165015
Title: A Phase 1, Multicenter, Parallel-Design, Single-Dose, Open-Label Study to Evaluate the Pharmacokinetics and Safety of LY3537031 in Participants With Normal Renal Function and Participants With Renal Impairment
Brief Title: A Study of Pharmacokinetics and Safety of LY3537031 in Participants With Normal Renal Function and Participants With Renal Impairment
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 27393; J2S-MC-GZMM (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Renal Impairment; Healthy; Renal Insufficiency; End Stage Renal Disease (ESRD)
MeSH Terms: conditions — Renal Insufficiency; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LY3537031 (Group 1) (Experimental): LY3537031 administered subcutaneously (SC) in a control group of participants with normal renal function
  Interventions: Drug: LY3537031
- LY3537031 (Groups 2-3) (Experimental): LY3537031 administered SC in groups of participants with impaired renal function
  Interventions: Drug: LY3537031
- LY3537031 (Group 3) (Experimental): LY3537031 administered SC in a group of participants with end-stage renal disease (ESRD) on hemodialysis
  Interventions: Drug: LY3537031

INTERVENTIONS:
Drug: LY3537031 — Administered SC

SUMMARY:
The purpose of this study is to assess the amount of LY3537031 that reaches the bloodstream and the time it takes for the body to get rid of it when given to participants with renal (kidney) impairment and to healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Have a body weight of 55 kilogram (kg) or more and body mass index (BMI) within the range 19.0 to 40.0 kilogram per square meter (kg/m²), inclusive
* Have no significant history of spontaneous or ethanol-induced hypoglycemia

Additional Inclusion Criteria for Healthy Participants in Control Group:

* Are healthy as determined by medical history, physical examination, and other screening procedures, with normal renal function, assessed by estimated glomerular filtration rate (eGFR) of at least 90 milliliter per minute (mL/min) at screening
* Have glycated hemoglobin (HbA1c) less than or equal to 6.5% at screening

Additional Inclusion Criteria for Participants with Severe Renal Impairment or with End-Stage Renal Disease (ESRD):

* Have stable severe renal impairment, assessed by eGFR less than 30 mL/min at screening, who have been on stable hemodialysis schedule for at least 3 months prior to planned dosing
* Have acceptable blood pressure and pulse rate
* If participants have Type 2 Diabetes Mellitus (T2DM), they must have a HbA1c equal to or less than 11.5% at the screening visit

Exclusion Criteria:

* Have a history of chronic liver disease, acute or chronic hepatitis, including a history of autoimmune hepatitis, any evidence for hepatic impairments
* Have a current, functional renal transplant. Non-functional renal allografts may be allowed
* Have a diagnosis or history of malignant disease within 5 years before screening (some exceptions are allowed)
* Have a family or personal history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome Type 2

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) of LY3537031 | Predose on day 1 up to week 8 post dose
  PK: AUC of LY3537031
PK: Maximum Concentration (Cmax) of LY3537031 | Predose on day 1 up to week 8 post dose
  PK: Cmax of LY3537031

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (3):
  - Omega Research Orlando LLC, Orlando, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Indiana University School of Medicine, Indianapolis, Indiana
- New Zealand Clinical Research Christchurch, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of Pharmacokinetics and Safety of LY3537031 in Participants With Normal Renal Function and Participants With Renal Impairment — https://trials.lilly.com/en-US/trial/650580